CLINICAL TRIAL: NCT03171402
Title: Astringency and Bitterness Perception Among High and Low Fruit and Vegetable Consumers
Brief Title: Astringency and Bitterness Perception
Status: Completed | Type: Observational
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Cordelia Running, PhD, Assistant Professor, Purdue University
Other Study IDs: 082-007
Record Dates: First submitted 2017-05-24; First posted 2017-05-31 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Taste Bitter-Salty

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low fruit and vegetable consumers: Participants with low F&V consumption, as defined by 24-hr dietary recall
  Interventions: Diagnostic Test: Astringency and bitterness perception
- High fruit and vegetable consumers: Participants with high F&V consumption, as defined by 24-hr dietary recall
  Interventions: Diagnostic Test: Astringency and bitterness perception

INTERVENTIONS:
Diagnostic Test: Astringency and bitterness perception — Participants will be involved in 1-4 experiments that test how they rate and differentiate between bitter and astringent flavored beverage samples

SUMMARY:
The investigators are conducting a study to better understand how the average consumer differentiates between bitter and astringent sensations, both of which are typically unpleasant sensations characteristic of some healthy foods. Astringency is the dry/rough sensation elicited by foods such as green bananas and some wines. Although trained scientists can differentiate between these stimuli, untrained participants rate them similarly, despite their differences. This confusion has created additional barriers in understanding the mechanism of astringent perception, which is currently debated. Understanding how to design experiments where untrained participants can clearly evaluate both sensations will lay the foundation to better understand astringency.

One mechanism that is believed to contribute to astringency is the interaction of astringent stimuli with salivary proteins. Interestingly, the salivary protein profile may be influenced by consumption of fruits and vegetables. Therefore, the investigators will evaluate how bitter and astringent perceptions differ among high and low consumers of fruits and vegetables by collecting saliva following exposure to the stimuli. This knowledge will inform approaches to increase the appeal of healthy food.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 18

Exclusion Criteria:

* issues with taste, smell, swallowing, choking, or salivation
* trying to gain or lose weight

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: * Not underweight (BMI > 18 kg/m^2)
  * Not be trying to gain or lose weight
  * Males and females 18-45
  * No known issues with taste, smell, swallowing, choking, or salivation
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2017-04-30 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Participant-generated sensory ratings of consumed samples | Through study completion, an average of three 30-minute visits
  Liking and flavor intensity ratings on the general labeled magnitude scale
Participant-generated groupings of consumed samples | Through study completion, an average of three 60-minute visits
  Hierarchical clustering of sample similarity
Participant-generated ratings of consumed samples relative to reference samples | Through study completion, an average of three 60-minute visits
  Similarity ratings of samples compared to three reference samples on a visual analog scale
Participant-generated "check-all-that-apply" ratings of consumed samples | Through study completion, an average of three 30-minute visits
  10-20 descriptors that are checked or unchecked by each participant to describe each sample

CONTACTS AND LOCATIONS:
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: No